CLINICAL TRIAL: NCT03913377
Title: Ocular Characteristics in Contact Lens and Spectacle Wear
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR-6332
Record Dates: First submitted 2019-04-10; First posted 2019-04-12 (Actual); Results first posted 2020-08-06 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-01

CONDITIONS: Visual Acuity
MeSH Terms: interventions — Eyeglasses

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Observational (Experimental): Eligible subjects that are habitual spectacle wearers will use their habitual optical correction and undergo ocular evaluations and questionnaires at the baseline and 1-week visit.
  Interventions: Device: Spectacles
- Interventional (Experimental): Eligible subjects that are habitual contact lens wearers who own spectacles will be randomized into 1 of 2 sequences (Spectacle/ACUVUE OASYS 1-Day or ACUVUE OASYS 1-Day/Spectacle)
  Interventions: Device: Spectacles; Device: ACUVUE OASYS®1-Day with HydraLuxe™ Technology

INTERVENTIONS:
Device: Spectacles — Subjects' own habitual spectacles
Device: ACUVUE OASYS®1-Day with HydraLuxe™ Technology — Test 1
  Arms: Interventional

SUMMARY:
This clinical study will investigate the difference in ocular characteristics between contact lens wear and spectacle wear among habitual contact lens wearers, using a 2-treatment by 2-period cross-over design. There will be a 1-week washout between the two study periods to eliminate any potential carryover effect.

ELIGIBILITY:
Inclusion Criteria:

* Potential subjects must satisfy all of the following criteria to be enrolled in the study:

  1. The subject will have completed the pre-screening Classification questionnaire.
  2. Subject must have a working cell phone capable of sending and receiving text messages.
  3. The subject must read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
  4. Appear able and willing to adhere to the instructions set forth in this clinical protocol.
  5. Between 18 and 42 (inclusive) years of age at the time of screening
  6. Be a current soft contact lens wearer in both eyes with a minimum of 5 days/week wear time over the last 1 month by self-report OR be a full-time spectacle wearer (7 days/ week) without contact lens wear over the last 6 months.
  7. Subjects must be willing to adhere to spectacle-only refractive correction for approximately 1 week.
  8. Subjects must possess a functional / usable pair of spectacles with which they can achieve 20/20 Snellen visual acuity or better at distance and near, and bring them to the visit
  9. The subject's vertex corrected spherical distance refraction must be in the range (+/-0.25 D) of -2.00 D to -6.00 D (inclusive) in each eye.
  10. The subject's vertex corrected refractive cylinder must be equal or less than -0.75 diopters in each eye.
  11. Contact lens wearers must have spherical best corrected visual acuity of 20/25 or better in each eye.
  12. Snellen visual acuity at distance and near must be within 1 line between subject's own spectacle and the manifest refraction, distance and near, OD & OS.

      Exclusion Criteria:
* Potential subjects who meet any of the following criteria will be excluded from participating in the study:

  1. Currently pregnant or lactating, by self-report
  2. Any ocular or systemic allergies, disease or use of medication which may interfere with contact lens wear and/or participation in the study (at the discretion of the investigator).
  3. Any active ocular abnormalities/conditions that may interfere with contact lens wear and/or participation in the study (at the discretion of the investigator).
  4. Any corneal distortion resulting from previous hard or rigid gas permeable contact lens wear
  5. Habitual contact lens wear modality as extended wear (≥1 night per month of extended wear).
  6. Habitual contact lens is rigid gas permeable, toric, monovision or multi-focal
  7. Habitual spectacle contains an add power, photochromic or tint.
  8. Any previous, or planned (during the course of the study) ocular surgery (e.g., radial keratotomy, PRK, LASIK, etc.)
  9. Participation in any contact lens or lens care product clinical trial within 2 weeks prior to study enrollment.
  10. Employee or employee's immediate family member of clinical site (e.g., Investigator, Coordinator, Technician)
  11. Current habitual use of Restasis, Xiidra, ocular steroids, or any medication (RX or OTC) that may interfere with contact lens wear and/or participation in the study (at the discretion of the investigator)
  12. Any ocular allergies, infections or other ocular abnormalities that are known to interfere with contact lens wear and/or participation in the study. This may include, but not be limited to entropion, ectropion, extrusions, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, aphakia, or corneal distortion.
  13. Any Grade 3 or greater biomicroscopy findings (this includes, corneal edema, corneal staining, corneal vascularization, conjunctival injection, tarsal abnormalities, bulbar injection) on the FDA classification scale (CTP-2018).
  14. Accommodative/binocular dysfunction, determined by study procedures.

Ages: 18 Years to 42 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2019-04-09 (Actual); Primary Completion 2019-06-14 (Actual); Study Completion 2019-06-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - VRC-East, Jacksonville, Florida
  - Sabal Eye Care, Longwood, Florida
  - Manhattan Vision Associates, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 78 subjects were enrolled into this study. Of those enrolled, 65 subjects were assigned to either the observational arm (21) or the interventional arm (44), while 13 subjects failed to meet all eligibility criteria.
Pre-assignment Details: Of the 21 subjects assigned to the observational arm, all subjects completed the study. Of the 44 subjects assigned to the interventional arm 2 subjects were discontinued. A total of 63 subjects completed the study.
Groups:
- Observational: Participants wearing their habitual spectacle wearers during the course of the study. This arm was included in the study to investigate ocular characteristics among habitual spectacle wearers which served as a reference group.
- Interventional: Test (Senofilcon A)/Control (Spectacle): Subjects randomized to this sequence received the Test lens (senofilcon A) during the first period and then worn their spectacles (Control) during the second period.
- Interventional: Control (Spectacle)/Test (Senofilcon A): Subjects randomized to this sequence worn their spectacles (Control) during the first period and then received the Test lens (senofilcon A) during the second period.
Period: Period 1
Arm/Group | Observational | Interventional: Test (Senofilcon A)/Control (Spectacle) | Interventional: Control (Spectacle)/Test (Senofilcon A)
Started | 21 | 22 | 22
Completed | 21 | 21 | 21
Not Completed | 0 | 1 | 1
Not completed — Test Article no longer available | 0 | 1 | 0
Not completed — No Longer Meets Eligibility Criteria | 0 | 0 | 1
Period: Period 2
Arm/Group | Observational | Interventional: Test (Senofilcon A)/Control (Spectacle) | Interventional: Control (Spectacle)/Test (Senofilcon A)
Started | 0 | 21 | 21
Completed | 0 | 21 | 21
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All subjects who were assigned either to the interventional arm or the observational arm based on their habitual vision corrections.
Groups:
- Observational Arm: Subjects wearing their habitual spectacle wearers during the course of the study. This arm was included in the study to investigate ocular characteristics among habitual spectacle wearers which served as a reference group.
- Interventional Arms: Participants assigned to the interentional arm to wear the Test lens and their own spectacles in a random order.
- Total: Total of all reporting groups
Arm/Group | Observational Arm | Interventional Arms | Total
Number analyzed (Participants) | 21 | 44 | 65
Age, Continuous [Mean (Standard Deviation); unit: Years] | 29.1 (6.40) | 28.9 (7.00) | 29.0 (6.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 26 | 42
  Male | 5 | 18 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 5 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 4 | 3 | 7
  White | 11 | 32 | 43
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 3 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 21 | 44 | 65

OUTCOME MEASURES:

1. Primary Outcome: Non-Invasive Break Up Time (NIBUT) or Non-Invasive Keratograph Break Up Time (NIKBUT)
Description: NIBUT/NIKBUT was measured as the time interval in seconds after the final blink to the first appearance of distortion in the reflected rings; or to the time that the participant has to blink due to discomfort. NIBUT is measured by a topographer (e.g. Medmont) via observation by the investigator and a stopwatch. NIKBUTis measured by the Oculus Keratograph and reported by the instrument. Different instrumentation was used depending on site availability. Combined measurements of pre-lens data collected for the interventional arm are reported. Only the interventional arm was reported since the primary analysis was conducted among habitual contact lens users. The average NIKBUT was reported for each treatment. Higher values indicate better performance
Time Frame: 1-Week Follow-up
Population: All subjects who had successfully completed all visits in the interventional arm and did not substantially deviate from the protocol.
Measure: Mean (Standard Deviation); unit: Seconds
Units Other Than Participants: eyes
Groups:
- Test (Senofilcon A): Subjects that wore the Test article in either the first or second period of the study.
- Control (Spectacle): Subjects that wore their spectacles in either the first or second period of the study.
Arm/Group | Test (Senofilcon A) | Control (Spectacle)
Number analyzed (Participants) | 41 | 41
Number analyzed (eyes) | 82 | 82
Seconds | 8.28 (4.482) | 11.10 (5.761)
Statistical Analysis 1: Comparison: Test (Senofilcon A) vs Control (Spectacle); The null and alternative hypotheses for testing significant difference between Test lens and Spectacles among habitual lens users with respect to NIBUT/NIKBUT; Test type: Equivalence — A statistically significant difference in NIBUT/NIKBUT between Test lens and Spectacles was concluded if the upper confidence limit of the 95% CI is below zero or the lower limit is above zero; Mixed Model Analysis; Kenward and Roger method was used for denominator degrees of freedom; LS Mean Difference = -2.79, 95% CI 2-sided [-4.14 to -1.44], Standard Error of Mean 0.678 — LS Mean difference was calculated as Test minus Control

2. Secondary Outcome: Total Scores of Meibomian Gland Expressibility (MGE)
Description: Meibomian gland expressiblity was assessed in three regions of the lower eyelid: temporal, central, and nasal. Each region is expressed and the overall grade of the region is evaluated using a four-grade scale: 0 = No Secretion, 1 = Inspissated, 2 = Colored/Cloudy Liquid, and 3 = Clear Liquid Oil. The total score was calculated as the sum of all grades across the three regions and ranged from 0 (no secretion) to 9, with higher scores indicating more MGE. Total scores were converted into a binary variable for the analysis purpose where Y=1 if the total score is greater than 6 and 0 otherwise. The percentage of participants with MGE total score greater than 6 was estimated. Only the interventional arm was reported since the secondary analysis was conducted among habitual contact lens users.
Time Frame: 1-Week Follow-up
Population: All participants who had successfully completed all visits in the interventional arm and did not substantially deviate from the protocol.
Measure: Mean (Standard Deviation); unit: Units on a scale
Units Other Than Participants: Eyes
Arm/Group | Test (Senofilcon A) | Control (Spectacle)
Number analyzed (Participants) | 41 | 41
Number analyzed (Eyes) | 82 | 82
Units on a scale | 8.5 (1.24) | 8.5 (1.28)
Statistical Analysis 1: Comparison: Test (Senofilcon A); Point estimates for Test and Control with 95% confidence intervals; Test type: Other — Estimated 95% confidence intervals for the point estimates of Test and Control; Mixed Model Analysis; Mean Proportion = 85.59, 95% CI 2-sided [43.2 to 97.89], Standard Error of Mean 1.038
Statistical Analysis 2: Comparison: Control (Spectacle); Point estimates for Test and Control with 95% confidence intervals; Test type: Other — Estimated 95% confidence intervals for the point estimates of Test and Control; Mixed Model Analysis; Mean Proportion = 84.17, 95% CI 2-sided [48.67 to 96.75], Standard Error of Mean 0.871

3. Secondary Outcome: Conjunctival Staining
Description: Conjunctival staining was graded and recorded by quadrant (Superior, Inferior, Nasal, and Temporal) using the following grading scale: Grade 0 = None, Grade 1 = Trace, Grade 2 = Mild, Grade 3 = Moderate, and Grade 4 = Severe. Average grade was calculated based on grades of the four quadrants. Only the interventional arm was reported since the secondary analysis was conducted among habitual contact lens users.
Time Frame: 1-Week Follow-up
Population: as for outcome 1
Measure: Number; unit: Number of Eyes
Units Other Than Participants: Eyes
Arm/Group | Test (Senofilcon A) | Control (Spectacle)
Number analyzed (Participants) | 41 | 41
Number analyzed (Eyes) | 82 | 82
Number of Eyes
  Nasal: Grade 0 | 41 | 59
  Nasal: Grade 1 | 34 | 23
  Nasal: Grade 2 | 7 | 0
  Nasal: Grade 3 | 0 | 0
  Nasal: Grade 4 | 0 | 0
  Temporal: Grade 0 | 55 | 79
  Temporal: Grade 1 | 25 | 3
  Temporal: Grade 2 | 2 | 0
  Temporal: Grade 3 | 0 | 0
  Temporal: Grade 4 | 0 | 0
  Inferior: Grade 0 | 40 | 75
  Inferior: Grade 1 | 34 | 6
  Inferior: Grade 2 | 7 | 1
  Inferior: Grade 3 | 1 | 0
  Inferior: Grade 4 | 0 | 0
  Superior: Grade 0 | 71 | 82
  Superior: Grade 1 | 9 | 0
  Superior: Grade 2 | 2 | 0
  Superior: Grade 3 | 0 | 0
  Superior: Grade 4 | 0 | 0
Statistical Analysis 1: Comparison: Test (Senofilcon A); Test type: Other — Estimated 95% confidence intervals for the point estimates of test; Mixed Model Analysis; Kenward and Rogers Metod was used for degrees of freedom; Mean = 0.52, 95% CI 2-sided [0.40 to 0.65], Standard Error of Mean 0.053; Point estimate was calculated for Test
Statistical Analysis 2: Comparison: Control (Spectacle); Test type: Other — Estimated 95% confidence intervals for the point estimates of Control; Mixed Model Analysis; Kenward and Rogers Metod was used for degrees of freedom; Mean = 0.13, 95% CI 2-sided [-0.19 to 0.44], Standard Error of Mean 0.036; Point estimates were calculated for Control

4. Secondary Outcome: Number of Eyes With Clinically Significant (Grade 3 or 4 of Overall Classification) Lid Wiper Epitheliopathy
Description: Horizontal lid margin staining and sagittal lid margin staining are graded for each eyelid (upper and lower) separately. The horizontal and sagittal grades are then averaged for each eyelid to obtain the upper lid average grade and lower lid average grade. The final grade is the average of the upper and lower lid average grades. Participants can be classified according to their final grades for each eye. The classification is defined as follows: "None" for final grades of 0, "Mild" for final grades between 0.25 and 1.00, "Moderate" for final grades between 1.25 and 2.00, and "Severe" for final graded between 2.25 and 3.00. Only the interventional arm was reported since the secondary analysis was planned to be conducted among habitual contact lens users only.
Time Frame: 1-Week Follow-up
Population: as for outcome 2
Measure: Number; unit: Number of eyes
Units Other Than Participants: Eyes
Arm/Group | Test (Senofilcon A) | Control (Spectacle)
Number analyzed (Participants) | 41 | 41
Number analyzed (Eyes) | 82 | 82
Number of eyes
  None | 36 | 31
  Mild | 15 | 19
  Moderate | 29 | 30
  Severe | 2 | 2
Statistical Analysis 1: Comparison: Test (Senofilcon A); Test type: Other — Estimated 95% confidence intervals for the point estimates of Test; Mixed Model Analysis; Mean Proportion = 30.7, 95% CI 2-sided [6.5 to 73.8], Standard Error of Mean 19.87 — Point estimates were calculated for Test
Statistical Analysis 2: Comparison: Control (Spectacle); Test type: Other — Estimated 95% confidence intervals for the point estimates of Control; Mixed Model Analysis; Mean Proportion = 27.9, 95% CI 2-sided [6.1 to 69.8], Standard Error of Mean 18.17 — Point estimates were calculated for Control

5. Secondary Outcome: Meibomian Gland Expressibility (MGE) Grades
Description: Meibomian gland expressiblity was assessed in three regions of the lower eyelid: temporal, central, and nasal. Each region is expressed and the overall grade of the region is evaluated using a four-grade scale: 0 = No Secretion, 1 = Inspissated, 2 = Colored/Cloudy Liquid, and 3 = Clear Liquid Oil. Only the interventional arm was reported since the secondary analysis was conducted among habitual contact lens users.
Time Frame: 1-Week Follow-up
Population: as for outcome 2
Measure: Number; unit: Units on a scale
Units Other Than Participants: Eyes
Arm/Group | Test (Senofilcon A) | Control (Spectacle)
Number analyzed (Participants) | 41 | 41
Number analyzed (Eyes) | 82 | 82
Units on a scale
  Central Lower Lid- Grade 0 | 0 | 0
  Central Lower Lid- Grade 1 | 0 | 0
  Central Lower Lid- Grade 2 | 10 | 6
  Central Lower Lid- Grade 3 | 72 | 76
  Nasal Lower Lid- Grade 0 | 0 | 1
  Nasal Lower Lid- Grade 1 | 2 | 0
  Nasal Lower Lid- Grade 2 | 9 | 7
  Nasal Lower Lid- Grade 3 | 71 | 74
  Temporal Lower Lid- Grade 0 | 2 | 6
  Temporal Lower Lid- Grade 1 | 4 | 2
  Temporal Lower Lid- Grade 2 | 5 | 5
  Temporal Lower Lid- Grade 3 | 71 | 69

ADVERSE EVENTS:
Time Frame: Throughout the duration of the study (about 3 weeks for subjects in the interventional arm and about 1 week for subjects in the observational arm).
Arm/Group | Observational | Test (Senofilcon A) | Control (Spectacle)
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/44 | 0/44
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/44 | 0/44
Other Adverse Events (participants affected / at risk) | 0/21 | 0/44 | 0/44

LIMITATIONS AND CAVEATS:
No study limitations were reported for this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-16): https://cdn.clinicaltrials.gov/large-docs/77/NCT03913377/Prot_SAP_000.pdf